CLINICAL TRIAL: NCT05511558
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Fosgonimeton (ATH-1017) Following a Single Subcutaneous Dose in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of [14C]-Fosgonimeton (ATH-1017)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry); Alturas Analytics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATH-1017-0102
Record Dates: First submitted 2022-08-15; First posted 2022-08-23 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosing Group (Experimental): All 8 subjects will receive a single dose of study drug
  Interventions: Drug: [14C]-Fosgonimeton

INTERVENTIONS:
Drug: [14C]-Fosgonimeton — Carbon-14 Radiolabeled Fosgonimeton
  Other Names: [14C]-ATH-1017

SUMMARY:
This is a Phase 1, open-label, nonrandomized, single-dose human, absorption, metabolism, and excretion study of [14C]-Fosgonimeton

DETAILED DESCRIPTION:
This is a Phase 1, open-label, nonrandomized, single-dose study, designed to evaluate the absorption, metabolism, and excretion of [14C]-Fosgonimeton. Healthy male subjects will receive a single subcutaneous dose of [14C]-Fosgonimeton.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 60 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by the investigator's discretion
4. Subjects and their partners will agree to use contraception during their participation
5. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

1. Significant history or clinical manifestation of any relevant, significant medical disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. Positive hepatitis panel and/or positive human immunodeficiency virus test.
4. Use or intend to use any prescription medications/products within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
5. Use or intend to use any nonprescription medications within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee).
6. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known) prior to dosing.
7. Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months
8. Poor peripheral venous access.
9. Subjects with exposure to significant diagnostic or therapeutic radiation (e.g., serial x-ray, computed tomography scan, barium meal)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Mass balance of total radioactivity from [14C]-Fosgonimeton | Samples collected pre-dose.
  Total radioactivity recovery (fet1-t2)
Mass balance of total radioactivity from [14C]-Fosgonimeton | Samples collected up to 9 days post-dose.
  Total radioactivity recovery (fet1-t2)
Routes/rates of elimination of [14C]-Fosgonimeton | Samples collected pre-dose.
  Total radioactivity recovery (fet1-t2) through routes of elimination (urine and feces).
Routes/rates of elimination of [14C]-Fosgonimeton | Samples collected up to 9 days post-dose.
  Total radioactivity recovery (fet1-t2) through routes of elimination (urine and feces).
Maximum observed plasma concentration (Cmax) of ATH-1017/ATH-1001 | Samples collected pre-dose and at predetermined timepoints within 24 hours post-dose.
  Cmax will be determined from plasma samples.
Time to maximum observed plasma concentration (Tmax) of ATH-1017/ATH-1001 | Samples collected pre-dose and at predetermined timepoints within 24 hours post-dose.
  Tmax will be determined from plasma samples
Area under the plasma concentration time curve (AUC) for of ATH-1017/ATH-1001 | Samples collected pre-dose and at predetermined timepoints within 24 hours post-dose.
  AUC will be determined from plasma samples.
Half-life (t1/2) of ATH-1017/ATH-1001 | Samples collected pre-dose and at predetermined timepoints within 24 hours post-dose.
  t1/2 will be determined from plasma samples.

SECONDARY OUTCOMES:
Quantitative metabolite profiles in plasma, urine, and feces after [14C]-Fosgonimeton administration | Samples collected pre-dose and at predetermined timepoints up to 9 days post-dose
  Quantification of ATH-1017 major metabolites in plasma and excreta.
The chemical structure of major metabolites in plasma, urine, and feces after [14C]-Fosgonimeton administration | Samples collected pre-dose and at predetermined timepoints up to 9 days post-dose
  Identification of ATH-1017 major metabolites in plasma (>10% relative total drug-related exposure) and excreta (>10% of excreted dose)
Incidence and severity of adverse events (safety and tolerability) of [14C]-Fosgonimeton when administered to healthy subjects | Samples collected pre-dose and at predetermined timepoints up to 17 days post-dose
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Madison, Wisconsin, United States